CLINICAL TRIAL: NCT02623595
Title: A Prospective Single-arm Multi-center Phase II Study: Assessment of the Safety and Abscopal Effects of SBRT in Combination With rhGM-CSF for Stage IV NSCLC Patients Who Failed in Second-line Chemotherapy
Brief Title: A Study of SBRT in Combination With rhGM-CSF for Stage IV NSCLC Patients Who Failed in Second-line Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient enrollment was hard mainly due to we need at least three lesions suitable for SBRT
Sponsor: Wuhan University (Other)
Collaborators: Tongji Hospital (Other); Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Conghua Xie,MD,PhD, Professor,MD,PhD,Director of Department of Radiation and Medical Oncology,Zhongnan Hospital, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHX-65
Record Dates: First submitted 2015-11-23; First posted 2015-12-07 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: non-small cell lung cancer; Granulocyte-Macrophage Colony-Stimulating Factor; Stereotactic body radiotherapy; abscopal effect; safety; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; regramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT+GM-CSF (Experimental): Metastasis lesion will be treated with a SBRT of 50Gy/5F from day 1 to day 5 in a cycle of 21 days.Subcutaneous injection of human recombined granulocyte-macrophage colony stimulating factor (125ug/m² per day) will be executed from day 1 to day 14 in this cycle. Another metastasis lesion will be treated likewise concurrently with rhGM-CSF in a consecutive cycle.
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: rhGM-CSF

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — A type of radiation therapy
  Other Names: SBRT; SABR
Drug: rhGM-CSF — Immune modulating agents
  Other Names: Recombined human granulocyte-macrophage colony stimulating factor

SUMMARY:
The purpose of this study is to determine whether stereotactic body radiotherapy (SBRT) combined with recombined human granulocyte-macrophage colony stimulating factor(rhGM-CSF) is safe, effective in the treatment of stage IV NSCLC patients who failed in second-line chemotherapy.

DETAILED DESCRIPTION:
Metastasis lesion will be treated with a SBRT of 50Gy/5F from day 1 to day 5 in one cycle.Subcutaneous injection of human recombined granulocyte-macrophage colony stimulating factor (125ug/m² per day) will be executed from day 1 to day 14 in this cycle. Another metastasis lesion will be treated likewise concurrently with rhGM-CSF in a consecutive cycle. Efficacy evaluation,especially abscopal effect evaluation, will be conducted at the end of therapy and every month after that. Adverse events will be recorded according to NCI-CTC version 4.03.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven non-small-cell lung cancer.
2. Stage IV according to UICC stage system(version 7,2009).
3. Progression after standard second-line chemotherapy.
4. At least Three evaluable lesions among which at least two must be suitable for SBRT.
5. ECOG performance status 0-2.
6. Expected lifespan ≥3 months.
7. Stable lab values:

   Hematological: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets ≥100×109/L, Hemoglobin ≥9 g/dL Renal: Creatinine OR Measured or calculated creatinine clearance (CrCl) (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≤1.5× the upper limit of normal (ULN) OR ≥60 mL/min for patient with creatinine levels >1.5× institutional ULN Hepatic: Total bilirubin ≤1.5×ULN OR Direct bilirubin ≤ULN for patients with total bilirubin levels >1.5×ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN OR ≤5×ULN for patients with liver metastases ,globulin≥20 g/L, albumin≥30 g/L.
8. Female subjects must have a negative urine or serum pregnancy test within 72 hours prior to taking study drug if of childbearing potential.
9. Able to understand and give written informed consent and comply with study procedures.

Exclusion criteria:

1. Any unstable systemic disease, including active infection, uncontrolled high blood pressure, unstable angina, newly observed angina pectoris within the past 3 months, congestive heart failure (New York heart association (NYHA) class II or higher), myocardial infarction onset six months before included into the group, and severe arrhythmia, liver, kidney, or metabolic disease in need of drug therapy.
2. Any clinical evidence suggests moderately severe chronic obstructive pulmonary disease (COPD) - [With COPD history or related risk factors, FEV1 / FVC < 70%, FEV1 < 80% estimated value, with or without chronic cough, sputum, dyspnea symptoms), active interstitial lung disease - ILD (FEV1 / FVC < 70%, FEV1 < 80% estimated value, carbon monoxide diffusion capacity in lung - DLCO < 40%, and high resolution CT (HRCT) confirmed as the diffuse pulmonary interstitial lesions] and other active pulmonary disease.
3. Previously diagnosed with autoimmune diseases, including but not limited to systemic lupus erythematous, rheumatoid arthritis, systemic vasculitis, scleroderma, dermatomyositis, autoimmune hemolytic anemia and autoimmune liver disease, autoimmune thyroiditis.
4. Human immunodeficiency virus (HIV) infection.
5. Women in pregnancy or lactation .
6. Medicine abusers(including alcohol, drugs or other addictive drugs abusers).
7. Patients with mental illness, considered as "can't fully understand the issues of this research".
8. Cancer history within 5 years apart from NSCLC before enrollment.
9. Histologically confirmed small cell carcinoma or other non NSCLC compositions in the cancer tissue.
10. Cancer treatment within 4 weeks, including but not limited to palliative surgery ,radiotherapy, chemotherapy and target therapy.
11. Tumor related immunotherapy within 1 year, including but not limited to immune cell therapy, tumor vaccine therapy, immune check-point monoclonal antibody related treatment, and cytokines treatment except for GM-CSF.
12. Allergy of rhGM-CSF and its accessories.
13. Contraindications to GM-CSF treatment.
14. Patients with unilateral lung.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2019-05 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
abscopal effect rate | at the time point of 4 weeks after completion of rhGM-CSF

SECONDARY OUTCOMES:
overall survival | 2 years
Incidence of Adverse events | 2 years
  All adverse events will be recorded
progression free survival | 2 years
objective response rate | 2 years
abscopal effect rate | at the time point of 2 months after completion of rhGM-CSF
Incidence of treatment-related adverse events | 2 years
  All treatment-related adverse events will be recorded
Incidence of immune-related adverse events | 2 years
  All Immune-related adverse events will be recorded

OTHER OUTCOMES:
Total T cells count in peripheral blood | pre-treatment,1, 2, 3, 6, 12 months after completion of rhGM-CSF
  To assess the absolute number of T cells in per milliliter peripheral blood pre- and post-therapy.
Absolute number of CD4+T, CD8+T and regulatory T cells | pre-treatment,1, 2, 3, 6, 12 months after completion of rhGM-CSF
  To assess ratio of effector T cells: regulatory T cells in per milliliter peripheral blood pre- and post-therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Conghua Xie, MD, PhD, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan hospital of Wuhan university, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Data of tumor response, abscopal effect rate and survival time will be available within 4 months of study completion

REFERENCES:
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Daly ME, Monjazeb AM, Kelly K. Clinical Trials Integrating Immunotherapy and Radiation for Non-Small-Cell Lung Cancer. J Thorac Oncol. 2015 Dec;10(12):1685-93. doi: 10.1097/JTO.0000000000000686. PMID 26484629
- [Background] Yokouchi H, Yamazaki K, Chamoto K, Kikuchi E, Shinagawa N, Oizumi S, Hommura F, Nishimura T, Nishimura M. Anti-OX40 monoclonal antibody therapy in combination with radiotherapy results in therapeutic antitumor immunity to murine lung cancer. Cancer Sci. 2008 Feb;99(2):361-7. doi: 10.1111/j.1349-7006.2007.00664.x. Epub 2008 Jan 14. PMID 18201271
- [Background] Slovin SF, Higano CS, Hamid O, Tejwani S, Harzstark A, Alumkal JJ, Scher HI, Chin K, Gagnier P, McHenry MB, Beer TM. Ipilimumab alone or in combination with radiotherapy in metastatic castration-resistant prostate cancer: results from an open-label, multicenter phase I/II study. Ann Oncol. 2013 Jul;24(7):1813-1821. doi: 10.1093/annonc/mdt107. Epub 2013 Mar 27. PMID 23535954
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Background] Younes E, Haas GP, Dezso B, Ali E, Maughan RL, Kukuruga MA, Montecillo E, Pontes JE, Hillman GG. Local tumor irradiation augments the response to IL-2 therapy in a murine renal adenocarcinoma. Cell Immunol. 1995 Oct 15;165(2):243-51. doi: 10.1006/cimm.1995.1211. PMID 7553889
- [Background] Golden EB, Demaria S, Schiff PB, Chachoua A, Formenti SC. An abscopal response to radiation and ipilimumab in a patient with metastatic non-small cell lung cancer. Cancer Immunol Res. 2013 Dec;1(6):365-72. doi: 10.1158/2326-6066.CIR-13-0115. PMID 24563870
- [Background] Hiniker SM, Chen DS, Reddy S, Chang DT, Jones JC, Mollick JA, Swetter SM, Knox SJ. A systemic complete response of metastatic melanoma to local radiation and immunotherapy. Transl Oncol. 2012 Dec;5(6):404-7. doi: 10.1593/tlo.12280. Epub 2012 Dec 1. PMID 23323154
- [Background] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785